CLINICAL TRIAL: NCT06648551
Title: Diagnostic Performance of CONUT as a Nutritional Screening Tool in Patients With Inflammatory Bowel Disease
Brief Title: Diagnostic Performance of Controlling Nutritional Status as a Nutritional Screening Tool in Patients With Inflammatory Bowel Disease
Acronym: CONUT
Status: Recruiting | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Nallely Bueno Hernández, Medical Sciences Researcher C, Hospital General de Mexico
Other Study IDs: DI/23/501/03/31
Record Dates: First submitted 2024-07-08; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Disease 5
MeSH Terms: conditions — Inflammatory Bowel Disease 5

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CONUT — It is a scale that uses albumin, lymphocytes, and cholesterol for the diagnosis of malnutrition

SUMMARY:
The objective of this observational study is to determine the diagnostic performance of CONUT as a nutritional screening tool in patients with Inflammatory Bowel Disease. The main questions to be answered are:

What is the sensitivity and specificity of CONUT as a nutritional screening tool in patients with Inflammatory Bowel Disease?

The participants will:

Undergo body composition analysis and a medical history review to understand the characteristics of their current condition, apply the GLIM criteria, and conduct their nutritional assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Gender unspecified
* Histologically confirmed Ulcerative Colitis
* Diagnosis confirmed by a specialist physician

Exclusion Criteria:

* Patients with any amputation or prosthesis
* Patients with a pacemaker
* Patients with any neoplasm
* Pregnancy or lactation
* With comorbidities such as diabetes, hypertension, heart failure, thyroid problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ulcerative Colitis patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Diagnostic test | one year
  sensitivity and specificity of CONUT as a nutritional screening tool in patients with Inflammatory Bowel Disease

CONTACTS AND LOCATIONS:
Locations (1):
- Nallely Hernandez Bueno, Mexico City, Cuauhtemoc, Mexico